CLINICAL TRIAL: NCT05170100
Title: Evaluating a Digital Intervention for Overactive Bladder: Protocol for a Single-arm, Multisite Pilot Clinical Trial
Brief Title: Evaluating a Digital Intervention for Overactive Bladder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Ireland, Galway, Ireland (Other)
Collaborators: Enterprise Ireland (Other Government)
Responsible Party: Principal Investigator, Emma Carr, Researcher, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CF20201467I
Record Dates: First submitted 2021-10-29; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NUIG OAB App (Experimental): Digital behaviour change intervention. Software-delivered intervention including best-practice behavioural therapy, and evidence-based dietetics, physiotherapy and psychology treatments to reduce the symptoms of overactive bladder.
  Interventions: Behavioral: NUIG OAB App

INTERVENTIONS:
Behavioral: NUIG OAB App — An interactive software-delivered 8-week intervention accessed through the patients' mobile device. It provides best-practice behavioural therapy, and delivers evidence-based dietetics, physiotherapy and psychology treatments to reduce the symptoms of overactive bladder.

SUMMARY:
Overactive Bladder is characterised by (I) Urgency: the sudden and compelling desire to pass urine with or without accidental leakage; (II) Frequency: the need to pass urine far more regularly than is considered normal; and (III) Nocturia: the need to pass urine several times during the night. This study aims to investigate the feasibility, acceptability and preliminary efficacy of a digital intervention (the NUIG OAB App) for overactive bladder. Furthermore, this study will help determine the most appropriate outcomes for use in the future definitive RCT and the effect size for future sample size calculations. Participants will complete an 8-week intervention designed to reduce the symptoms of OAB, delivered through the NUIG OAB App. Participants will be asked to complete online surveys at baseline, 4 weeks and 8 weeks and an in-app Bladder Diary at weeks 1 and 8. There will be no in-person contact with participants by the study team.

ELIGIBILITY:
Inclusion Criteria:

1. On waiting list for Urogynaecologist at participating hospital
2. Referred for Overactive bladder from GP
3. Symptoms of Overactive bladder to include at least one of the following: urgency of urination, frequency of urination or urge incontinence.
4. Female
5. 18 years or older
6. Own a smartphone

Exclusion Criteria:

1. Active/Recurrent urinary tract infection
2. Urinary retention
3. Bladder Pain Syndrome/ interstitial cystitis
4. Pelvic/gynae cancer
5. Pregnant
6. Dementia
7. Kidney problems
8. Stroke
9. Have/had a neuro-stimulation implant for treatment of OAB

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2021-11-07 (Actual)

PRIMARY OUTCOMES:
Change in International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life Module (ICIQ-OABqol) | baseline and week 8
  Change from baseline patient-reported overactive bladder related quality of life at week 8. Minimum score 25, maximum score 160. Greater values indicating increased impact on quality of life
Change in International Consultation on Incontinence Questionnaire Overactive Bladder Module (ICIQ-OAB) | baseline and week 8
  Change from baseline patient-reported overactive bladder symptoms at week 8. Minimum score 0, maximum score 16. Greater values indicate increased symptom severity.
Change in Digital Bladder Diary frequency of urination | baseline & week 8
  Change from baseline frequency of urination at week 8.
  Frequency of urination measured in-app, in real-time as number of urinations per day logged by user for 3 days at baseline and 3 days in week 8.

SECONDARY OUTCOMES:
Programme adherence | data collected throughout the 8 week intervention.
  Total number of seconds spent on app from day 1 of week 1 to day 7 of week 8. Total number of times app accessed between day 1 of week 1 and day 7 of week 8. Total number of in-app 'challenges' completed throughout the 8 week intervention.
Mobile Applications Rating Scale, user version (MARSu) | week 4
  User reported ratings of app quality based on Engagement, Functionality, Aesthetics, and Information. Minimum score 20, maximum score 100. Greater values indicate higher app quality.
Patient Global impression of improvement | week 8
  One item questionnaire with Likert scale of 1 to 7. Greater values indicate disimproved condion.
Change in International Consultation on Incontinence Questionnaire Overactive Bladder Quality of Life Module (ICIQ-OABqol) | baseline and week 4
  Change from baseline patient-reported overactive bladder related quality of life at week 4. Minimum score 25, maximum score 160. Greater values indicate increased impact on quality of life.
Change in International Consultation on Incontinence Questionnaire Overactive Bladder Module (ICIQ-OAB) | baseline and week 4
  Change from baseline patient-reported overactive bladder symptoms at week 4. Minimum score 0, maximum score 16. Greater values indicate increased symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Staunton, Principal Investigator — National University of Ireland, Galway
Locations (3):
- Ireland (3):
  - The Rotunda Hospital, Dublin
  - The National Maternity Hospital, Dublin
  - Galway University Hospital, Galway

IPD SHARING:
Plan to Share IPD: No